CLINICAL TRIAL: NCT07061444
Title: Effects of Different Inspiratory Muscle Training Protocols in Hematopoietic Stem Cell Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ceren Derya Gültekin (Other)
Responsible Party: Sponsor-Investigator, Ceren Derya Gültekin, Ceren Derya Gültekin, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24-207
Record Dates: First submitted 2024-12-31; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Hematopoietic Stem Cell Transplantation (HSCT); Pulmonary Rehabilitation; Inspiratory Muscle Training
Keywords: inspiratory muscle training; pulmonary rehabilitation; hematopoietic stem cell transplantation; respiratory therapy; respiratory muscle

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Inspiratory Muscle Training Group (Active Comparator): Fifteen patients meeting the inclusion criteria will undergo standard inspiratory muscle training using the PowerBreathe Classic device (HaB International Ltd., Southam, UK). IMT will be performed at 40% of the maximum inspiratory pressure (MIP), with weekly re-assessment of MIP by the responsible researcher to adjust the training workload. Each session will consist of 8-10 diaphragmatic breaths, followed by a rest interval of 5-10 seconds, lasting 15 minutes per session. Training will be conducted twice daily, five days per week.
  Vital signs, including heart rate and oxygen saturation, will be monitored continuously throughout the exercises, and measurements will also be taken before, after, and during the first minute of recovery. This progressive IMT protocol aims to optimize inspiratory muscle strength through evidence-based threshold pressure loading, ensuring patient safety and effective respiratory muscle adaptation over time.
  Interventions: Other: Inspiratory Muscle Training
- 2. Functional Inspiratory Muscle Training Group (Active Comparator): Fifteen patients will undergo functional respiratory muscle training integrating inspiratory muscle training (IMT) and functional exercises. The POWERbreathe IMT device, using a threshold loading technique, will be set at 40% of maximum inspiratory pressure (MIP) and adjusted weekly based on updated MIP values. Training sessions will be conducted face-to-face, three times per week, for 30 minutes under physiotherapist supervision, while classical IMT will continue on other days. During each session, heart rate, oxygen saturation, fatigue, and dyspnoea perception will be monitored before, during, and after exercises, including the first minute of recovery. The six-week program will involve progressive functional exercises classified into three difficulty levels-easy, medium, and hard-spanning two-week intervals. Patients will be instructed to inhale through the POWERbreathe device during movement and exhale upon returning to the starting position.
  Interventions: Other: Functional Inspiratory Muscle Training
- 3. Control Group (Placebo Comparator): Sham protocol will be applied to 15 randomly selected patients. All vital signs of the patient will be taken before and after exercise training and during the 1st minute recovery period. Oxygen saturation monitoring and heart rate will be measured throughout the exercise. Type: threshold loading inspiratory muscle training (PowerBreath classic will be used.) Progression: will be studied at 10% of the re-measured MIP at the beginning of each week.
  Interventions: Other: Sham Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — Inspiratory muscle training will be performed at 40% of MIP workload, 1 set of 8-10 diaphragmatic respirations for 15 minutes, with 5-10 seconds rest intervals between sets. 5 days a week, 2 sessions per day.
  Arms: 1. Inspiratory Muscle Training Group
Other: Functional Inspiratory Muscle Training — This study investigates the integration of functional inspiratory muscle training (IMT) with conventional physiotherapy. Patients will perform inspiratory muscle training using the threshold loading technique with the POWERbreathe IMT device, combined with functional exercises. The functional IMT protocol will be administered face-to-face, 3 days a week, for 30 minutes per session over a 6-week period. Resistance on the IMT device will be set to 40% of the patient's maximal inspiratory pressure (MIP) and adjusted weekly based on measured MIP values. Exercises will be categorized into three progressive difficulty levels (easy, medium, and hard), with each stage lasting 2 weeks. Patients will inhale through the POWERbreathe IMT device during exercise movements and exhale during the return phase, ensuring simultaneous respiratory muscle activation and functional training.
  Arms: 2. Functional Inspiratory Muscle Training Group
Other: Sham Inspiratory Muscle Training — Control group will be performed at 10% of the MIP workload, 1 set of 8-10 diaphragmatic breaths for 15 minutes, with 5-10 seconds rest intervals between sets. 2 sessions per day, 5 days a week.
  Arms: 3. Control Group

SUMMARY:
Introduction: After haematopoietic stem cell transplantation (HSCT), patients often experience complications such as respiratory difficulties, fatigue and decreased quality of life.

The aim of the study was to compare the effectiveness of different inspiratory muscle training (IMT) protocols on respiratory muscle strength and endurance, dyspnoea, maximal exercise capacity, diaphragmatic function, respiratory function parameters, peripheral muscle strength, fatigue, quality of life, oxidative stress parameters, muscle biomarkers and inflammatory biomarkers in HSCT recipients during the transplantation process.

Method: The study will include patients between 18-65 years of age, who are able to walk and understand the instructions, who do not have orthopedic, neurological or cardiac disorders and who will undergo haematopoietic stem cell transplantation. Patients with cognitive impairments; orthopedic or neurological diseases that may affect the evaluation of physical fitness tests; patients with comorbidities such as asthma, COPD will not be included in the study. In cases where the exercise group subjects' attendance to the training protocol is interrupted for 3 sessions or more consecutively, the voluntariness to participate in the research is lost during the research process, and clinical haemodynamic instability develops in the subjects, the participant will be excluded from the study. Patients in whom exercise training is contraindicated such as acute bleeding, haemoglobin value <5 g/dl, platelet count ≤10000 mm3, high fever (body temperature >38◦C), severe pain, confusion, dizziness, nausea and vomiting will not be included in the exercise.

It is planned as a prospective, randomised controlled and single blinded study. Triple blinding could not be performed due to the executive's evaluation and implementation of the study protocol. Patients included in the study will be randomly divided into 3 study groups of 15 people each. Stratified randomisation technique will be used. A total of 45 haematopoietic stem cell transplant patients will be included in the study. Patients will be evaluated 3 times: before exercise therapy (pre-HSCT), before and after starting the preparatory regime and after exercise therapy (post-HSCT). Primary assessment measures are dyspnoea, maximal exercise capacity, respiratory muscle strength and endurance, diaphragmatic respiration, oxidative stress parameters, inflammatory markers, muscle biomarkers, pulmonary function test. Secondary assessment measures were peripheral muscle strength, fatigue, depression, and quality of life.

The research arms consisted of a total of 45(15;15;15) people in 3 groups: 'standard inspiratory muscle training group', 'functional respiratory muscle training group' and 'control group' with 15 people in each group. All patients in the control and research groups will receive inspiratory muscle training for a total of 30 minutes twice a day, every weekday during the transplantation period, starting at the end of the session in which their initial assessment was made. Functional respiratory muscle training group will perform functional exercises simultaneously with inspiratory muscle training 3 days a week (Monday-Wednesday-Friday or Tuesday-Thursday-Saturday). All exercises will be supervised by a physiotherapist.

The most important originality of this study is that it is the first study to investigate the effects of functional respiratory muscle training on respiratory parameters, diaphragm function, peripheral muscle strength, maximum oxygen consumption, dyspnoea, fatigue, depression and quality of life in HSCT recipients. It is the first randomised controlled study to demonstrate the effect of inspiratory muscle training on diaphragmatic function in HSCT recipients and it is one of the rare studies in which exercise capacity will be evaluated by cardiopulmonary exercise test. It is also the first study to examine the relationship between inspiratory muscle training and muscle biomarkers and oxidative stress parameters in HSCT recipients.

H0: There is no difference in the effectiveness of different inspiratory muscle training protocols on maximal exercise capacity, respiratory muscle strength, respiratory muscle endurance, diaphragmatic function, oxidative stress parameters, muscle biomarkers, inflammatory biomarkers, dyspnoea, peripheral muscle strength, quality of life, fatigue, depression in haematopoietic stem cell transplant recipients.

H1: There is a difference in the effectiveness of different inspiratory muscle training protocols on maximal exercise capacity, respiratory muscle strength, respiratory muscle endurance, diaphragmatic function, oxidative stress parameters, muscle biomarkers, inflammatory biomarkers, dyspnoea, peripheral muscle strength, quality of life, fatigue, depression in haematopoietic stem cell transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Planned haematopoietic stem cell transplantation in the adult bone marrow transplant unit
* Between the ages of 18-65
* Under standard medical treatment, including immunosuppressives, antibiotics and other medications
* Ability to walk, co-operate and be clinically stable
* No history of orthopaedic, neurological, cardiac disorders

Exclusion Criteria:

* Cognitive disorders
* Have orthopaedic or neurological diseases that may affect the assessment of physical fitness tests
* Having comorbidities such as asthma, COPD
* Conditions in which exercise training is contraindicated, such as acute bleeding, haemoglobin value <5 g/dl, platelet count ≤10000 mm3, high fever (body temperature >38◦C), severe pain, confusion, dizziness, nausea and vomiting
* Patients with pneumonia or any acute infection

  -≥ 3 consecutive sessions of interruption of the exercise group subjects' attendance to the training protocol
* Loss of willingness to participate in the research during the research process
* Development of clinical haemodynamic instability in patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-02 (Estimated); Primary Completion 2026-08-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Dyspnea Perception Measurement | "Through study completion, an average of 1 year"
  Dyspnea perception will be assessed using the Modified Borg Scale and the Modified Medical Research Council (MMRC) Dyspnea Scale.
  Modified Borg Scale: A subjective scale to assess dyspnea at rest and/or during activity. The scale ranges from 0-10, where 0 indicates no dyspnea and 10 indicates very severe dyspnea, reflecting the participant's perceived breathlessness.
  Modified MMRC Dyspnea Scale: This scale evaluates dyspnea during daily activities. It is graded as follows:
  0: No dyspnea except for severe activity.
  1. Dyspnea during fast walking or uphill climbing.
  2. Dyspnea causes slower movement or stops on flat ground.
  3. Dyspnea causes stopping after walking 100 meters or a few minutes.
  4. Dyspnea occurs during dressing or undressing, preventing leaving the house.
  Unit of Measure:
  Modified Borg Scale: 0-10 points
  MMRC Dyspnea Scale: Grade 0-4
Cardiopulmonary Function Measurement | "Through study completion, an average of 1 year"
  Cardiopulmonary function will be assessed using the Cardiopulmonary Exercise Test (CPET) with the MES VO₂max Finder device (Poland), providing measurements of VO₂, VCO₂, VE, RER, and ventilatory threshold following ATS and ERS standards.
  Protocol:
  Pre-test Preparation: Avoid caffeine and vigorous exercise for 24 hours prior.
  Test Protocol: The Modified Bruce protocol with progressive increases in speed (2.7 to 8.8 km/h) and incline (0 to 20%) every 3 minutes.
  Vital Signs Monitoring: Heart rate, blood pressure, SpO₂, dyspnea, and fatigue monitored.
  Test Duration: 8-12 minutes, ending when two criteria are met (exhaustion, 90% max heart rate, RER ≥ 1.10, or blood lactate > 8.0 mmol/L).
  Cooldown: 3-minute cooldown post-test.
  Gas exchange analyzed breath-by-breath, with calibration per ATS/ERS guidelines.
  Unit of Measure:
  VO₂: mL/min VCO₂: mL/min VE: L/min RER: Ratio Ventilatory Threshold: L/min
Respiratory Muscle Strength Measurement | "Through study completion, an average of 1 year"
  Respiratory muscle strength will be assessed by measuring Maximum Inspiratory Pressure (MIP) and Maximum Expiratory Pressure (MEP) using the Micro Medical Micro RPM device (Rochester, UK), with measurements recorded in cmH₂O.
  MIP: Measured during maximal inspiration against a closed airway after full expiration.
  MEP: Measured during maximal expiration against a closed airway after full inspiration.
  Both MIP and MEP will be maintained for 1-3 seconds. Three measurements will be taken, and the best value will be recorded. Results will be expressed as a percentage of normal reference values adjusted for age and gender.
  Disposable, personalized mouthpieces and filters will be used to prevent infection, following ERS (2019) guidelines.
  Unit of Measure:
  MIP and MEP: cmH₂O, expressed as a percentage of normal reference values.
Respiratory Muscle Endurance Measurement | "Through study completion, an average of 1 year"
  Respiratory muscle endurance will be assessed using the Powerbreath Plus MR (HaB International Ltd., Southam, England), an inspiratory muscle training device employing a constant threshold load technique. The resistance of the device will be set at 60% of the participant's Maximum Inspiratory Pressure (MIP) value.
  During the test:
  The device will be placed in the participant's mouth, and the nose will be closed with a clip.
  The participant will be instructed to breathe through the device for a maximum of 10 minutes.
  Participants will be informed before the test that they can remove the device and stop the test if they feel excessive shortness of breath or discomfort.
  The time the participant is able to continue the test will be recorded in seconds.
  Unit of Measure:
  The unit of measure for this outcome is seconds for the duration the participant can continue the test.
Diaphragm Function and Thickness Measurement | "Through study completion, an average of 1 year"
  Diaphragm function and thickness will be assessed using Aplio XG ultrasonography (Toshiba, Japan) with patients in a supine position.
  Diaphragm Thickness: Measured using B-mode ultrasound with a 7 MHz transducer at the 9th intercostal space on the anterior axillary line at the end of expiration. Left hemidiaphragm imaging will not be performed due to anatomical limitations.
  Diaphragm Movement: Analyzed using M-mode ultrasonography with a 3.5 MHz transducer in a longitudinal semi-coronal plane. Excursion during calm breathing, deep breathing, and sniff test excursion will be assessed. The difference in diaphragm movement between inspiration and expiration will be calculated across three respiratory cycles.
  Unit of Measure:
  Diaphragm thickness and excursion will be expressed in millimeters (mm).
Inflammatory Markers Measurement | "Through study completion, an average of 1 year"
  Blood samples will be collected in blood collection tubes and centrifuged at 3,000 x g for 10 minutes to obtain the serum supernatant. The serum samples will be stored at -80°C until the day of the experiment.
  The following inflammatory markers will be measured:
  Proinflammatory markers: TNF-α and IL-6
  Anti-inflammatory markers: IL-2 and IL-10
  These markers will be measured using commercially available ELISA-based kits (Mybiosource Co., USA).
  Unit of Measure:
  The unit of measure will be expressed in pg/mL or ng/mL, depending on the kit's specifications for each marker.
Oxidative Stress Parameters Measurement | "Through study completion, an average of 1 year"
  Blood samples will be collected in blood collection tubes, centrifuged at 3,000 x g for 10 minutes to obtain serum supernatant, and stored at -80°C until analysis.
  Total Antioxidant Status (TAS): Measured by spectrophotometry (Thermo Scientific, Varioskan LUX, USA) using a commercial kit (Rel Assay Diagnostics, Turkey). Antioxidants reduce the ABTS radical to its colorless form, with absorbance at 660 nm correlating to TAS.
  Total Oxidant Status (TOS): Measured using a commercial kit (Rel Assay Diagnostics, Turkey) and spectrophotometrically (Thermo Scientific, Varioskan LUX, USA).
  Unit of Measure:
  TAS: mmol Trolox Equiv/L
  TOS: µmol H₂O₂ Equiv/L (or as per the kit specifications)
Muscle Biomarkers Measurement | "Through study completion, an average of 1 year"
  Serum CK-MM and CK-MB concentrations will be measured using ELISA-based commercial kits. Microwells pre-coated with monoclonal antibodies will capture the biomarkers, followed by detection using a biotin-conjugated antibody. After washing, HRP-conjugated avidin will be added, and TMB substrate will be used for colorimetric detection. Absorbance will be measured at 450 nm using a spectrophotometric plate reader (Thermo Scientific, USA).
  Blood samples (15 mL × 3 tubes) will be collected twice, before and after treatment, in gel biochemistry tubes at İstinye University laboratories. Serum will be obtained by centrifugation and stored at -80°C until analysis. In addition, CRP, hemoglobin, platelet, and albumin levels will be recorded from patient follow-up files.
  Unit of Measure:
  CK-MM and CK-MB concentrations: ng/mL (as per the ELISA kit specifications)
Pulmonary Function Test | "Through study completion, an average of 1 year"
  The pulmonary function test will be performed using a spirometer (Cosmed Pony FX, Italy) following ATS/ERS guidelines. The test will measure:
  Forced Vital Capacity (FVC)
  Forced Expiratory Volume in the First Second (FEV1)
  FEV1/FVC ratio
  Peak Expiratory Flow (PEF)
  Forced Expiratory Midflow Rate (FEF25-75%)
  The test will be conducted in a sitting position, with the best of three technically acceptable maneuvers demonstrating 95% agreement selected for analysis. Parameters will be expressed as a percentage of predicted values adjusted for age, height, and gender. Sterilization procedures, disposable, and personalized mouthpieces/filters will be used to prevent infection.
  Unit of Measure:
  FVC, FEV1, FEV1/FVC, PEF, FEF25-75%: Percentage of predicted values (adjusted for age, height, and gender)

SECONDARY OUTCOMES:
Peripheral Muscle Strength Measurement | "Through study completion, an average of 1 year"
  Peripheral muscle strength will be assessed using a portable manual muscle strength measuring device (Model 01165, Lafayette, IN, USA) and a Jamar Hydraulic Hand Dynamometer (Jamar, Nottinghamshire, UK). The muscles assessed include:
  Upper extremity: Shoulder abductor, shoulder flexor, elbow flexor, and elbow extensor.
  Lower extremity: Hip flexor and knee extensor.
  Grip strength will be measured in a sitting position with the elbow flexed at 90° and wrist neutral. Three measurements will be taken for each side (right and left), and the best value recorded in kilograms (kg) for grip strength and Newton-meters (Nm) for knee extensor strength. The measurements will be interpreted using reference equations from Andrews et al.
  Unit of Measure:
  Grip strength: kg Knee extensor strength: Nm
  Minimal Clinical Significance:
  Knee extensor strength: 17.2 Nm
  Grip strength: 6.25 kg
Fatigue Perception Measurement | "Through study completion, an average of 1 year"
  Fatigue perception will be assessed using the Turkish adaptation of the Fatigue Severity Scale (FSS). The self-administered scale consists of nine items that evaluate the severity of fatigue experienced by the participant. Each item is rated on a 7-point scale, where 1 indicates "strongly disagree" and 7 indicates "strongly agree."
  The total score can range from a minimum of 9 to a maximum of 63. A total score of 36 or above indicates severe fatigue according to the criteria established by Armutlu et al. (2007).
  The scale provides a reliable assessment of the participant's perceived fatigue severity, allowing for the evaluation of changes over time.
Depression Measurement | "Through study completion, an average of 1 year"
  Depression will be assessed using the 21-item self-administered Beck Depression Inventory (BDI), developed by Beck et al. The scale consists of 21 items that assess depression-specific conditions. Each item is scored on a 4-point scale, where scores range from 0 to 3. A higher score indicates a higher level of depression.
  The total score on the inventory can range from 0 (no depression) to 63 (severe depression). A score above 17 is accepted as indicative of the presence of depression.
  The unit of measure for this outcome is the total score, reported in points.
Quality of Life Measurement | "Through study completion, an average of 1 year"
  Quality of life will be assessed using the Turkish adaptation of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30, Version 3.0). The Turkish version has been proven to be reliable and valid for use with patients. The questionnaire consists of 30 items, designed to evaluate the quality of life of cancer patients. It comprises nine subscales, which include:
  Five functional scales: Physical, role, cognitive, emotional, and social functioning.
  One global health and quality of life scale.
  Three symptom scales: Fatigue, nausea and vomiting, pain, dyspnoea, sleep disturbance, loss of appetite, constipation, diarrhoea, and financial difficulties.
  Additionally, the questionnaire includes items assessing the financial impact of the disease and its treatment.
  The unit of measure for this outcome is the total score, reported in points, derived from responses to the individual items within the subscales.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plans to share individual participant data.